CLINICAL TRIAL: NCT04819516
Title: A Single-arm, Single-center Exploratory Study of the Safety and Effectiveness of High-intensity Focused Ultrasound Therapy Combined With REGOTORI for Metastatic Colorectal Cancer
Brief Title: Study of the Safety and Effectiveness of HIFU Combined With REGOTORI for Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Ying Yuan, MD, Professor, Department of Medical Oncology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFUREGONIVO2101
Record Dates: First submitted 2021-01-27; First posted 2021-03-29 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Extracorporeal Shockwave Therapy; toripalimab; regorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HIFU with REGOTORI (Experimental)
  Interventions: Procedure: high-intensity focused ultrasound therapy; Drug: Toripalimab

INTERVENTIONS:
Procedure: high-intensity focused ultrasound therapy — Patients will receive high-intensity focused ultrasound therapy in local site.
Drug: Toripalimab — Toripalimab plus regorafenib
  Other Names: Regorafenib

SUMMARY:
This study intends to perform high-intensity focused ultrasound combined with REGOTORI in patients with multiline drug-resistant metastatic colorectal cancer to explore the safety and efficacy of patients. Patients receive HIFU local treatment combined with REGOTORI treatment, and receive corresponding clinical data collection at different follow-up points, including necessary data from various laboratories, CT/MRI, and immune function tests that are exactly the same as before surgery collection.

ELIGIBILITY:
Inclusion Criteria:

* The subject has metastatic colorectal cancer, and the first and second-line standard treatments have failed
* There is at least one target lesion that can be treated with HIFU
* Voluntarily accept this treatment clinical research, and sign the "Subject Informed Consent"
* 18-75 years old, no gender limit
* The level of physical strength of the Eastern Cooperative Oncology Group (ECOG): PS<=2
* The expected survival time is greater than 3 months
* No chemotherapy or radiotherapy within 21 days before enrollment
* The function of major organs is basically normal

Exclusion Criteria:

* Pregnant or lactating women
* People infected with HIV, hepatitis C virus and Treponema pallidum
* There is an active infection that requires systemic treatment (such as active tuberculosis)
* Severe infection within 4 weeks before starting the study treatment
* Subjects who have received allogeneic tissue/solid organ transplantation
* The patient suffers from major vascular disease or irregular bleeding disease
* Suffer from physiological or pathological malnutrition diseases, chronic diarrhea, cachexia, etc.
* The patient has autoimmune diseases, such as (but not limited to) multiple sclerosis, systemic lupus erythematosus and inflammatory bowel disease, vitiligo
* The patient has a history of serious drug or food allergy (for example, allergy to protein)
* The patient has serious heart disease (including but not limited to: myocardial infarction, cardiomyopathy, valvular disease, malignant arrhythmia, etc.), severe liver and kidney damage, uncontrolled blood sugar and blood pressure (the subject's blood pressure, After using antihypertensive drugs, it still cannot be controlled within the normal range; fasting blood glucose is still >10mmol/L after using antihypertensive drugs)
* The patient has uncontrollable seizures or loss of insight due to mental illness
* In the 12 months before screening, the patient has a history of drug abuse, drug abuse, and long-term alcoholism
* Within 3 months before screening, the patient is participating in other clinical studies
* Other situations that cannot participate in clinical research.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-12-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse events | 3 months from baseline
Adverse events | 6 months from baseline
Adverse events | 9 months from baseline
Adverse events | 12 months from baseline
Number of Participants With Abnormal Laboratory Values | 3 months from baseline
Number of Participants With Abnormal Laboratory Values | 6 months from baseline
Number of Participants With Abnormal Laboratory Values | 9 months from baseline
Number of Participants With Abnormal Laboratory Values | 12 months from baseline

SECONDARY OUTCOMES:
Number of Participants With Abnormal Tumor markers | 12 months from baseline
Number of Participants With Abnormal Tumor markers | 3 months from baseline
Number of Participants With Abnormal Tumor markers | 6 months from baseline
Number of Participants With Abnormal Tumor markers | 9 months from baseline
Disease Control Rate | From Baseline to primary completion date, about 60 months
Progression Free Survival | From Baseline to primary completion date, about 60 months
QoL | 12 months from baseline
  Quality of life is assessed using the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30. It will be evaluated at Screening, Tumor Assessment Visit and End of Treatment visit.
Numeric rating scale | 12 months from baseline
  Numerical Rating Scale (pain measurement) minimum: 0, means no pain maximum: 10, means unbearable physical pain

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, Ph.D & MD, Study Chair — The Second Affiliated Hospital of Medical College of Zhejiang University
Locations (1):
- the Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang, China